CLINICAL TRIAL: NCT01197300
Title: A 1-year, Multicenter, Open-label Extension to CZOL446H2337 to Evaluate Safety and Efficacy of Zoledronic Acid Twice Yearly in Osteoporotic Children Treated With Glucocorticoids
Brief Title: 1 Year Open-label Extension to CZOL446H2337 Safety and Efficacy Trial of Zoledronic Acid Twice Yearly in Osteoporotic Children Treated With Glucocorticoids
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CZOL446H2337E1; 2010-020399-41 (EudraCT Number)
Record Dates: First submitted 2010-09-07; First posted 2010-09-09 (Estimated); Results first posted 2019-09-20 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-08

CONDITIONS: Osteoporosis
Keywords: Osteoporosis, children and adolescents, zoledronic acid, chronic inflammation, Duchenne muscular dystrophy, glucocorticoids, chronic inflammatory conditions
MeSH Terms: conditions — Osteoporosis; Muscular Dystrophy, Duchenne | interventions — Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Zoledronic acid (Experimental): Twice yearly 0.05 mg/kg (max 5 mg) i.v infusion (at least 30 minutes) of zoledronic acid
  Interventions: Drug: Zoledronic acid

INTERVENTIONS:
Drug: Zoledronic acid — intravenous infusion

SUMMARY:
This 1-year open-label extension to CZOL446H2337 is designed to evaluate the safety and efficacy of zoledronic acid twice yearly in osteoporotic children treated with glucocorticoids.

ELIGIBILITY:
Key Inclusion criteria:

Written informed consent before any study-related procedure.

Group 1:

1. Children and adolescents, male or female, 6-19 years old, who met the inclusion criteria for entry into the Core study and who took at least one dose of study drug and have completed Visit 8 of the CZOL446H2337 Core study.
2. Patient must be enrolled into the extension at Visit 9 up to 10 months after Visit 5 (month 6) of the Core study.
3. Patients who followed the regimen of calcium and vitamin D intake as required in the Core study through diet or supplementation.

Group 2:

1. Children and adolescents, male or female, 5 - 17 years old who met the inclusion criteria for entry into the Core study but were not enrolled because of clinically significant back pain from vertebral fracture and the preexisting clinical care at the Investigator site is to treat this type of patient with a bisphosphonate.
2. Confirmed diagnosis of non-malignant conditions (including but not limited to rheumatic conditions, inflammatory bowel disease, Duchenne muscular dystrophy, nephrotic syndrome), treated with systemic glucocorticoids (i.v. or oral) within the 12 months preceding enrollment in the study (any duration)
3. LS-BMD Z-score of -0.5 or worse confirmed by the central imaging vendor
4. Evidence of at least 1 vertebral compression fracture (at least Genant Grade 1 vertebral compression or radiographic signs of vertebral compression) confirmed by central reading OR At least one lower OR 2 upper extremity long-bone, low-trauma, fracture which occurred sometime within the 2 years or preceding enrollment in the study, confirmed by radiological report. (*Low trauma fracture is defined as falling from standing height or less).

Key Exclusion criteria:

1. Major protocol violation in the Core Study (Group 1 only).
2. Prior use of bisphosphonates (Group 2 only) or sodium fluoride (doses for osteoporosis not for dental hygiene).
3. Hypocalcemia and hypophosphatemia: any value (age-matched) below the normal range at Visit 8 or 8A.
4. Vitamin D deficiency (serum 25-hydroxy vitamin D concentrations of < 20 ng/mL or < 50 nmol/L) at Visit 8 (Group 1) or Visit 8A (Group 2).
5. Renal impairment defined as an estimated glomerular filtration rate (GFR) < 60 mL/min/1.73 m2 at screening based on the Schwartz formula at Visit 8 or 8 A; a serum creatinine above the normal range at Visit 9 (Group 1) or an increase between Visit 8A and Visit 9 greater than 0.5 mg/dL (44.2 μmol/L) for Group 2.
6. Female patients of child bearing potential are eligible only if they are not pregnant/non-lactating. Females of child bearing potential must be practicing a medically acceptable form of birth control for greater than 2 months prior to screening visit and consent to pregnancy tests during the study.

Ages: 5 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2010-10-25 (Actual); Primary Completion 2019-02-27 (Actual); Study Completion 2019-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (9):
- Novartis Investigative Site, Westmead, New South Wales, Australia
- Canada (3):
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Montreal, Quebec
- Novartis Investigative Site, Budapest, Hungary
- Russia (2):
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Saint Petersburg
- Novartis Investigative Site, Soweto, Gauteng, South Africa
- Novartis Investigative Site, West Midlands, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Background] Black DM, Delmas PD, Eastell R, Reid IR, Boonen S, Cauley JA, Cosman F, Lakatos P, Leung PC, Man Z, Mautalen C, Mesenbrink P, Hu H, Caminis J, Tong K, Rosario-Jansen T, Krasnow J, Hue TF, Sellmeyer D, Eriksen EF, Cummings SR; HORIZON Pivotal Fracture Trial. Once-yearly zoledronic acid for treatment of postmenopausal osteoporosis. N Engl J Med. 2007 May 3;356(18):1809-22. doi: 10.1056/NEJMoa067312. PMID 17476007
- [Background] Glorieux FH, Bishop NJ, Plotkin H, Chabot G, Lanoue G, Travers R. Cyclic administration of pamidronate in children with severe osteogenesis imperfecta. N Engl J Med. 1998 Oct 1;339(14):947-52. doi: 10.1056/NEJM199810013391402. PMID 9753709
- [Background] Plotkin LI, Weinstein RS, Parfitt AM, Roberson PK, Manolagas SC, Bellido T. Prevention of osteocyte and osteoblast apoptosis by bisphosphonates and calcitonin. J Clin Invest. 1999 Nov;104(10):1363-74. doi: 10.1172/JCI6800. PMID 10562298
- [Background] Reid IR, Brown JP, Burckhardt P, Horowitz Z, Richardson P, Trechsel U, Widmer A, Devogelaer JP, Kaufman JM, Jaeger P, Body JJ, Brandi ML, Broell J, Di Micco R, Genazzani AR, Felsenberg D, Happ J, Hooper MJ, Ittner J, Leb G, Mallmin H, Murray T, Ortolani S, Rubinacci A, Saaf M, Samsioe G, Verbruggen L, Meunier PJ. Intravenous zoledronic acid in postmenopausal women with low bone mineral density. N Engl J Med. 2002 Feb 28;346(9):653-61. doi: 10.1056/NEJMoa011807. PMID 11870242
- [Background] Ward L, Tricco AC, Phuong P, Cranney A, Barrowman N, Gaboury I, Rauch F, Tugwell P, Moher D. Bisphosphonate therapy for children and adolescents with secondary osteoporosis. Cochrane Database Syst Rev. 2007 Oct 17;2007(4):CD005324. doi: 10.1002/14651858.CD005324.pub2. PMID 17943849

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in 10 centers in 6 countries: Australia (1), Canada (4), Hungary (1), United Kingdom (1), Russian Federation (2), and South Africa (1).
Pre-assignment Details: This was an open label extension to the Core study CZOL446H2337 (NCT00799266), where all patients received zoledronic acid. However, the study groups from the Core study were used to compare the patient populations within this extension phase, who received the same treatment under each particular group.
Groups:
- Core Treatment Zoledronic Acid; Core Treatment: Placebo: Twice yearly 0.05 mg/kg (max 5 mg) i.v infusion (at least 30 minutes) of zoledronic acid
Period: Overall Study
Arm/Group | Core Treatment Zoledronic Acid | Core Treatment: Placebo
Started (All enrolled patients were included in the Full Analysis Set (FAS) and Safety Set) | 10 | 15
Completed | 10 | 13
Not Completed | 0 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Core Treatment Zoledronic Acid | Core Treatment: Placebo | Total
Number analyzed (Participants) | 10 | 15 | 25
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age at extension informed consent
  Years | 15.3 (2.58) | 13.2 (3.38) | 14.0 (3.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 7 | 10 | 17
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 8 | 13 | 21
  Black | 2 | 1 | 3
  Native American | 0 | 1 | 1
Lumbar Spine Bone Mineral Density (BMD) Z-score [Mean (Standard Deviation); unit: Z-score] — Lumbar Spine Bone Mineral Density (BMD) Z-score in the Full Analysis (FAS) population. Extension baseline was defined as the last non-missing measurement on or prior to the date of first study drug infusion in the extension study. Bone mass, as measured by DXA, is reported as BMC (g) or areal BMD (g/cm2). These values are compared with reference values from healthy youth of similar age, sex, and race/ ethnicity to calculate a z score, the number of SDs from the expected mean. A BMC or BMD z score that is >2 SDs below expected (< -2.0) is referred to as "low for age".
  Z-score | -1.568 (1.0196) | -2.291 (1.0712) | -2.002 (1.0909)
Lumbar Spine Bone Mineral Content (BMC) [Mean (Standard Deviation); unit: gram (g)] — Lumbar Spine Bone Mineral Content (BMC) in the Full Analysis (FAS) population. Extension baseline was defined as the last non-missing measurement on or prior to the date of first study drug infusion in the extension study.
  gram (g) | 42.106 (15.6967) | 25.890 (7.3089) | 32.376 (13.7584)
Total body Bone Mineral Content (BMC) [Mean (Standard Deviation); unit: gram (g)] — Total body Bone Mineral Content (BMC) in the Full Analysis (FAS) population. Extension baseline was defined as the last non-missing measurement on or prior to the date of first study drug infusion in the extension study. Population: All patients with non-missing assessment
  gram (g)
    number analyzed (Participants) | 9 | 13 | 22
    (all) | 1976.698 (636.2144) | 1144.613 (253.5405) | 1485.011 (605.2026)
Serum Procollagen type 1 amino-terminal propeptide (P1NP) [Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)] — Serum Procollagen type 1 amino-terminal propeptide (P1NP) in the Full Analysis (FAS) population. Extension baseline was defined as the last non-missing measurement on or prior to the date of first study drug infusion in the extension study.
  nanogram per milliliter (ng/mL) | 141.300 (100.8111) | 523.933 (475.5547) | 370.880 (415.1329)
Bone specific alkaline phosphatase (BSAP) [Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)] — Serum Bone specific alkaline phosphatase (BSAP) in the Full Analysis (FAS) population. Extension baseline was defined as the last non-missing measurement on or prior to the date of first study drug infusion in the extension study.
  nanogram per milliliter (ng/mL) | 25.841 (14.8595) | 49.737 (36.6580) | 40.179 (31.7718)
Serum Cross linked N-telopeptide (NTX) [Mean (Standard Deviation); unit: nmol BCE/L] — Serum Cross linked N-telopeptide (NTX) in the Full Analysis (FAS) population. Extension baseline was defined as the last non-missing measurement on or prior to the date of first study drug infusion in the extension study.
  nmol BCE/L | 19.092 (8.3760) | 42.217 (25.2275) | 35.967 (24.3991)
Serum Tartrate-resistant acid phosphatase isoform 5b (TRAP-5b) [Mean (Standard Deviation); unit: U/L] — Serum Tartrate-resistant acid phosphatase isoform 5b (TRAP-5b) in the Full Analysis (FAS) population. Extension baseline was defined as the last non-missing measurement on or prior to the date of first study drug infusion in the extension study.
  U/L | 5.338 (2.5097) | 8.636 (5.2925) | 7.316 (4.6283)
Second metacarpal cortical width [Mean (Standard Deviation); unit: millimeter (mm)] — Second metacarpal cortical width in the Full Analysis (FAS) population. Metacarpal cortical width of "0" was not included. An analysis of covariance model used with treatment, pooled centers, underlying condition treated with glucocorticoids at baseline value as explanatory variables and pooled centers as random effect. Population: All patients with non-missing assessment
  millimeter (mm)
    number analyzed (Participants) | 8 | 13 | 21
    (all) | 0.45 (0.207) | 0.38 (0.163) | 0.41 (0.179)

OUTCOME MEASURES:

1. Primary Outcome: Long-term Safety of Zoledronic Acid for the Treatment of Osteoporotic Children Treated With Glucocorticoids.
Description: Analysis of absolute and relative frequencies for treatment emergent Adverse Event (AE), Serious Adverse Event (SAE) and Deaths by primary System Organ Class (SOC) to demonstrate that zoledronic acid given long-term, over an additional 12 months from the Core study (CZOL446H2337), is safe for the treatment of osteoporotic children treated with glucocorticoids through the monitoring of relevant clinical and laboratory safety parameters.
Time Frame: Baseline 1 (Visit 1 of the Core Study) through Month 24 (Visit 15/Final Extension Visit)
Population: The Safety population, which consisted of all patients who had been exposed to at least one infusion of study drug, was considered.
Measure: Count of Participants; unit: Participants
Arm/Group | Core Treatment Zoledronic Acid | Core Treatment: Placebo
Number analyzed (Participants) | 10 | 15
Participants
  On-treatment Adverse Events (AEs) | 7 | 12
  On-treatment Serious Adverse Events (SAEs) | 3 | 0
  On-treatment Deaths | 0 | 0

2. Secondary Outcome: Mean Change From Baseline 1 (Visit 1 of the Core Study) in Lumbar Spine Bone Mineral Density (BMD) Z-score at Month 18 and 24 by Core Treatment Group.
Description: Lumbar Spine Bone Mineral Density (BMD) Z-score was determined by the central imaging vendor at the final visit of Core study (Visit 8) or at 1st infusion visit (Visit 9), and thereafter at Visit 12 (Month 18) and Visit 15 (Month 24) (final Extension Study visit/EOS) of Extension study. The methods to be used to measure Lumbar Spine BMD Z-score were described in the respective DXA Manuals provided by central imaging vendor. Positive changes from Core baseline indicated an improvement in condition.
Time Frame: Month 18 (Visit 12 of the Extension Study), Month 24 (Visit 15/Final Extension Visit)
Population: The Full Analysis population, which consisted of all randomized patients who had both Core Baseline and at least one post-baseline lumbar spine BMD Z-score in the Extension study, was considered.
Measure: Least Squares Mean (Standard Error); unit: Z-score
Arm/Group | Core Treatment Zoledronic Acid | Core Treatment: Placebo
Number analyzed (Participants) | 10 | 15
Z-score
  Lumbar Spine BMD Z-score Change at Month 18: number analyzed (Participants) | 10 | 13
  Lumbar Spine BMD Z-score Change at Month 18 | -40.648 (14.1205) | -44.348 (14.0348)
  Lumbar Spine BMD Z-score Change at Month 24: number analyzed (Participants) | 10 | 14
  Lumbar Spine BMD Z-score Change at Month 24 | -46.161 (12.4486) | -67.913 (12.1722)
Statistical Analysis 1: Comparison: Core Treatment Zoledronic Acid vs Core Treatment: Placebo; Lumbar Spine BMD Z-score Change at Month 18; Test type: Superiority — Difference in least squares mean = LS mean for the Core treatment Zoledronic acid group - LS mean for the Core treatment Placebo group; p = 0.8505, ANCOVA — An analysis of covariance (ANCOVA) model was performed with Core treatment, pooled centers, underlying condition treated with GCs and Core baseline lumbar spine BMD Z-score as explanatory variables and pooled centers as random effect; Difference in LS mean = 3.700, 95% CI 2-sided [-37.242 to 44.642]
Statistical Analysis 2: Comparison: Core Treatment Zoledronic Acid vs Core Treatment: Placebo; Lumbar Spine BMD Z-score Change at Month 24; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.2180, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Difference in LS mean = 21.752, 95% CI 2-sided [-14.126 to 57.630]

3. Secondary Outcome: Mean Change From Baseline 1 (Visit 1 of the Core Study) in Lumbar Spine Bone Mineral Content (BMC) at Month 18 and 24 by Core Treatment Group.
Description: Lumbar Spine Bone Mineral Content (BMC) was determined by the central imaging vendor at the final visit of Core study (Visit 8) or at 1st infusion visit (Visit 9), and thereafter at Visit 12 (Month 18) and Visit 15 (Month 24) (final Extension Study visit/EOS) of Extension study. The methods to be used to measure BMC were described in the respective DXA Manuals. Positive changes from Core baseline indicated an improvement in condition.
Time Frame: Month 18 (Visit 12 of the Extension Study), Month 24 (Visit 15/Final Extension Visit)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: gram
Arm/Group | Core Treatment Zoledronic Acid | Core Treatment: Placebo
Number analyzed (Participants) | 10 | 15
gram
  Lumbar Spine BMC Change at Month 18: number analyzed (Participants) | 10 | 13
  Lumbar Spine BMC Change at Month 18 | 12.293 (1.7749) | 9.933 (1.6717)
  Lumbar Spine BMC Change at Month 24: number analyzed (Participants) | 10 | 13
  Lumbar Spine BMC Change at Month 24 | 15.845 (2.2217) | 14.666 (2.0500)
Statistical Analysis 1: Comparison: Core Treatment Zoledronic Acid vs Core Treatment: Placebo; Lumbar Spine BMC Change at Month 18; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.3544, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Difference in LS mean = 2.360, 95% CI 2-sided [-2.886 to 7.606]
Statistical Analysis 2: Comparison: Core Treatment Zoledronic Acid vs Core Treatment: Placebo; Lumbar Spine BMC Change at Month 24; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.7050, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Difference in LS mean = 1.179, 95% CI 2-sided [-5.281 to 7.639]

4. Secondary Outcome: Mean Change From Baseline 1 (Visit 1 of the Core Study) in Total Body BMC at Month 18 and 24 by Core Treatment Group.
Description: Total body BMC were determined by the central imaging vendor at the final visit of Core study (Visit 8) or at 1st infusion visit (Visit 9), and thereafter at Visit 12 (Month 18) and Visit 15 (Month 24) (final Extension Study visit/EOS) of Extension study. The methods to be used to measure BMC were described in the respective DXA Manuals. Positive changes from Core baseline indicated an improvement in condition.
Time Frame: Month 18 (Visit 12 of the Extension Study), Month 24 (Visit 15/Final Extension Visit)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: gram
Arm/Group | Core Treatment Zoledronic Acid | Core Treatment: Placebo
Number analyzed (Participants) | 10 | 15
gram
  Total body BMC Change at Month 18: number analyzed (Participants) | 8 | 10
  Total body BMC Change at Month 18 | 387.721 (87396.2756) | 266.592 (87396.2698)
  Total body BMC Change at Month 24: number analyzed (Participants) | 9 | 11
  Total body BMC Change at Month 24 | 496.997 (120.9281) | 431.323 (123.5462)
Statistical Analysis 1: Comparison: Core Treatment Zoledronic Acid vs Core Treatment: Placebo; Total body BMC Change at Month 18; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.5310, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Difference in LS mean = 121.129, 95% CI 2-sided [-291.000 to 533.258]
Statistical Analysis 2: Comparison: Core Treatment Zoledronic Acid vs Core Treatment: Placebo; Total body BMC Change at Month 24; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.7347, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Difference in LS mean = 65.674, 95% CI 2-sided [-344.067 to 475.415]

5. Secondary Outcome: Mean Change From Baseline 1 (Visit 1 of the Core Study) in Serum P1NP at Month 18 and 24 by Core Treatment Group.
Description: Serum Procollagen type 1 amino-terminal propeptide (P1NP) was collected at the final visit Core study at Visit 8, or at 1st infusion visit (Visit 9), and thereafter at Visit 12 (Month 18) and Visit 15 (Month 24) (final Extension study Visit/EOS) of Extension study according to the instructions provided in the Laboratory Manual. The samples were analyzed in batches at the laboratory. Decrease or negative changes from Core baseline indicated a pharmacological response to therapy.
Time Frame: Month 18 (Visit 12 of the Extension Study), Month 24 (Visit 15/Final Extension Visit)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: nanogram per milliliter (ng/mL)
Arm/Group | Core Treatment Zoledronic Acid | Core Treatment: Placebo
Number analyzed (Participants) | 10 | 15
nanogram per milliliter (ng/mL)
  Serum P1NP Change at Month 18: number analyzed (Participants) | 10 | 12
  Serum P1NP Change at Month 18 | -169.837 (86.8640) | -22.157 (82.6761)
  Serum P1NP Change at Month 24: number analyzed (Participants) | 10 | 13
  Serum P1NP Change at Month 24 | -228.068 (54.1402) | -95.631 (53.0765)
Statistical Analysis 1: Comparison: Core Treatment Zoledronic Acid vs Core Treatment: Placebo; Serum P1NP Change at Month 18; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.4143, ANCOVA — An analysis of covariance (ANCOVA) model was performed on the transformed data with Core treatment, pooled centers, underlying condition treated with glucocorticoids and loge as explanatory variables and pooled centers as random effect; The transformed data was calculated by dividing the post-baseline value by the baseline value and then applying the loge transformation; Difference in LS mean = -147.680, 95% CI 2-sided [-394.410 to 99.049]
Statistical Analysis 2: Comparison: Core Treatment Zoledronic Acid vs Core Treatment: Placebo; Serum P1NP Change at Month 24; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.1266, ANCOVA — [p-value comment as in outcome 5, analysis 1]; [statistical method as in outcome 5, analysis 1]; Difference in LS mean = -132.437, 95% CI 2-sided [-286.452 to 21.579]

6. Secondary Outcome: Mean Change From Baseline 1 (Visit 1 of the Core Study) in BSAP at Month 18 and 24 by Core Treatment Group.
Description: Bone specific alkaline phosphatase (BSAP) was collected at the final visit Core study at Visit 8, or at 1st infusion visit (Visit 9), and thereafter at Visit 12 (Month 18) and Visit 15 (Month 24) (final Extension study Visit/EOS) of Extension study according to the instructions provided in the Laboratory Manual. The samples were analyzed in batches at the laboratory. Decrease or negative changes from Core baseline indicated a pharmacological response to therapy.
Time Frame: Month 18 (Visit 12 of the Extension Study), Month 24 (Visit 15/Final Extension Visit)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: nanogram per milliliter (ng/mL)
Arm/Group | Core Treatment Zoledronic Acid | Core Treatment: Placebo
Number analyzed (Participants) | 10 | 15
nanogram per milliliter (ng/mL)
  BSAP Change at Month 18: number analyzed (Participants) | 10 | 12
  BSAP Change at Month 18 | -13.716 (8.5909) | 3.975 (8.0523)
  BSAP Change at Month 24: number analyzed (Participants) | 10 | 13
  BSAP Change at Month 24 | -9.675 (6.4159) | -6.013 (5.9316)
Statistical Analysis 1: Comparison: Core Treatment Zoledronic Acid vs Core Treatment: Placebo; BSAP Change at Month 18; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.2123, ANCOVA — [p-value comment as in outcome 5, analysis 1]; [statistical method as in outcome 5, analysis 1]; Difference in LS mean = -17.691, 95% CI 2-sided [-41.925 to 6.543]
Statistical Analysis 2: Comparison: Core Treatment Zoledronic Acid vs Core Treatment: Placebo; BSAP Change at Month 24; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.4852, ANCOVA — [p-value comment as in outcome 5, analysis 1]; [statistical method as in outcome 5, analysis 1]; Difference in LS mean = -3.662, 95% CI 2-sided [-21.479 to 14.155]

7. Secondary Outcome: Mean Change From Baseline 1 (Visit 1 of the Core Study) in Serum NTX at Month 18 and 24 by Core Treatment Group.
Description: Serum Cross linked N-telopeptide (NTX) was collected at the final visit Core study at Visit 8, or at 1st infusion visit (Visit 9), and thereafter at Visit 12 (Month 18) and Visit 15 (Month 24) (final Extension study Visit/EOS) of Extension study according to the instructions provided in the Laboratory Manual. The samples were analyzed in batches at the laboratory. Decrease or negative changes from Core baseline indicated a pharmacological response to therapy.
Time Frame: Month 18 (Visit 12 of the Extension Study), Month 24 (Visit 15/Final Extension Visit)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: nmol BCE/L
Arm/Group | Core Treatment Zoledronic Acid | Core Treatment: Placebo
Number analyzed (Participants) | 10 | 15
nmol BCE/L
  Serum NTX Change at Month 18: number analyzed (Participants) | 9 | 10
  Serum NTX Change at Month 18 | -17.577 (168.8975) | -12.916 (168.8965)
  Serum NTX Change at Month 24: number analyzed (Participants) | 9 | 14
  Serum NTX Change at Month 24 | -17.450 (2.3585) | -14.891 (2.0590)
Statistical Analysis 1: Comparison: Core Treatment Zoledronic Acid vs Core Treatment: Placebo; Serum NTX Change at Month 18; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.9009, ANCOVA — [p-value comment as in outcome 5, analysis 1]; [statistical method as in outcome 5, analysis 1]; Difference in LS mean = -4.661, 95% CI 2-sided [-16.647 to 7.325]
Statistical Analysis 2: Comparison: Core Treatment Zoledronic Acid vs Core Treatment: Placebo; Serum NTX Change at Month 24; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.9472, ANCOVA — [p-value comment as in outcome 5, analysis 1]; [statistical method as in outcome 5, analysis 1]; Difference in LS mean = -2.558, 95% CI 2-sided [-8.864 to 3.747]

8. Secondary Outcome: Mean Change From Baseline 1 (Visit 1 of the Core Study) in Serum TRAP-5b at Month 18 and 24 by Core Treatment Group.
Description: Serum Tartrate-resistant acid phosphatase isoform 5b (TRAP 5b) were collected at the final visit Core study at Visit 8, or at 1st infusion visit (Visit 9), and thereafter at Visit 12 (Month 18) and Visit 15 (Month 24) (final Extension study Visit/EOS) of Extension study according to the instructions provided in the Laboratory Manual. The samples were analyzed in batches at the laboratory. Decrease or negative changes from Core baseline indicated a pharmacological response to therapy. Decrease or negative changes from Core baseline indicated a pharmacological response to therapy.
Time Frame: Month 18 (Visit 12 of the Extension Study), Month 24 (Visit 15/Final Extension Visit)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: U/L
Arm/Group | Core Treatment Zoledronic Acid | Core Treatment: Placebo
Number analyzed (Participants) | 10 | 15
U/L
  Serum TRAP-5b Change at Month 18: number analyzed (Participants) | 10 | 12
  Serum TRAP-5b Change at Month 18 | -2.661 (0.8126) | -1.179 (0.7725)
  Serum TRAP-5b Change at Month 24: number analyzed (Participants) | 10 | 13
  Serum TRAP-5b Change at Month 24 | -2.670 (0.7158) | -2.260 (0.6701)
Statistical Analysis 1: Comparison: Core Treatment Zoledronic Acid vs Core Treatment: Placebo; Serum TRAP-5b Change at Month 18; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.4600, ANCOVA — [p-value comment as in outcome 5, analysis 1]; [statistical method as in outcome 5, analysis 1]; Difference in LS mean = -1.482, 95% CI 2-sided [-3.805 to 0.841]
Statistical Analysis 2: Comparison: Core Treatment Zoledronic Acid vs Core Treatment: Placebo; Serum TRAP-5b Change at Month 24; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.9236, ANCOVA — [p-value comment as in outcome 5, analysis 1]; [statistical method as in outcome 5, analysis 1]; Difference in LS mean = -0.410, 95% CI 2-sided [-2.423 to 1.603]

9. Secondary Outcome: Number of Participants With New Vertebral Fractures During the 12 Month Extension Period by Core Treatment Group.
Description: New vertebral fractures are defined as fractures of Genant grade 1 or higher that occur at lumbar or thoracic spine from first extension dose infusion to the end of the study in a previously normal vertebra.
Time Frame: Month 24 (Visit 15/Final Extension Visit)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Core Treatment Zoledronic Acid | Core Treatment: Placebo
Number analyzed (Participants) | 10 | 15
Participants | 1 | 1
Statistical Analysis 1: Comparison: Core Treatment Zoledronic Acid vs Core Treatment: Placebo; New vertebral fractures at Month 12 Extension; Test type: Other — The number and percentage of patients with new vertebral fractures during the 12 month Extension period was presented by Core treatment group. Between-treatment differences were evaluated using Fisher's exact test; p = 1.0000, Fisher Exact

10. Secondary Outcome: Number of Participants With New Morphometric Vertebral Fractures During the 12 Month Extension Period by Core Treatment Group.
Description: Vertebral morphometry (or concave index) was calculated using the average ratio between mid-height and posterior height from L1 to L4 and performed by a central reader. A new morphometric vertebral fractures during the 12 month Extension Period was defined as a morphometric vertebral fracture present at Month 24 X-ray which was not present at the Extension Baseline (Baseline 2).
Time Frame: Month 24 (Visit 15/Final Extension Visit)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Core Treatment Zoledronic Acid | Core Treatment: Placebo
Number analyzed (Participants) | 10 | 15
Participants | 1 | 1
Statistical Analysis 1: Comparison: Core Treatment Zoledronic Acid vs Core Treatment: Placebo; New morphometric vertebral fractures at Month 12 Extension; Test type: Other — The number and percentage of patients with new morphometric vertebral fractures during the 12 month extension period was presented by core treatment group. Between-treatment differences will be evaluated using Fisher's exact test; p = 1.0000, Fisher Exact

11. Secondary Outcome: Percentage of Patients With Reduction in Pain From Baseline 1 (Visit 1 of the Core Study) at Month 15, 18, 21 and 24 by Core Treatment Group.
Description: Pain was evaluated at each visit (at office and telephone visit) at the final visit of the Core study and first visit of the Extension study (Visit 9), Visits 11 (Month 15), 12 (Month 18), 14 (Month 21) and 15 (Month 24) using the Faces Pain Scale-Revised (FPS-R). Children were selecting the face that best fits their pain. The pain score ranged from 0 (No Pain) to 10 (Very Much Pain). The reduction in pain from Core baseline by visit was evaluated based on whether or not patients had a decrease in their FPS-R from baseline. If pain remained the same or worsened from baseline a patient was classified as '0' and if the pain scale decreased then the patient was classified as '1'.
Time Frame: Month 15, Month 18, Month 21, Month 24
Population: as for outcome 2
Measure: Number; unit: Percentage of Patients
Arm/Group | Core Treatment Zoledronic Acid | Core Treatment: Placebo
Number analyzed (Participants) | 10 | 15
Percentage of Patients
  Reduction in Pain at Month 15: number analyzed (Participants) | 9 | 13
  Reduction in Pain at Month 15 | 55.6 | 46.2
  Reduction in Pain at Month 18: number analyzed (Participants) | 10 | 12
  Reduction in Pain at Month 18 | 30.0 | 50.0
  Reduction in Pain at Month 21: number analyzed (Participants) | 10 | 12
  Reduction in Pain at Month 21 | 30.0 | 50.0
  Reduction in Pain at Month 24: number analyzed (Participants) | 10 | 13
  Reduction in Pain at Month 24 | 30.0 | 38.5
Statistical Analysis 1: Comparison: Core Treatment Zoledronic Acid vs Core Treatment: Placebo; Reduction in Pain at Month 15; Test type: Other; p = 0.3971, Regression, Logistic — Presented by treatment group and evaluated using a logistic regression model with Core treatment, pooled centers, underlying condition treated with glucocorticoids and Core baseline pain score as explanatory variables; Odds Ratio (OR) = 4.73, 95% CI 2-sided [0.13 to 173.07]
Statistical Analysis 2: Comparison: Core Treatment Zoledronic Acid vs Core Treatment: Placebo; Reduction in Pain at Month 18; Test type: Other; p = 0.6046, Regression, Logistic — [p-value comment as in outcome 11, analysis 1]; Odds Ratio (OR) = 0.01, 95% CI 2-sided [0.01 to 999.99]
Statistical Analysis 3: Comparison: Core Treatment Zoledronic Acid vs Core Treatment: Placebo; Reduction in Pain at Month 21; Test type: Other; p = 0.6046, Regression, Logistic — [p-value comment as in outcome 11, analysis 1]; Odds Ratio (OR) = 0.01, 95% CI 2-sided [0.01 to 999.99]
Statistical Analysis 4: Comparison: Core Treatment Zoledronic Acid vs Core Treatment: Placebo; Reduction in Pain at Month 24; Test type: Other; p = 0.8750, Regression, Logistic — [p-value comment as in outcome 11, analysis 1]; Odds Ratio (OR) = 1.31, 95% CI 2-sided [0.05 to 38.04]

12. Secondary Outcome: Mean Change From Baseline (Core and Extension) in 2nd Metacarpal Cortical Width at Month 24 by Core Treatment Group.
Description: Left postero-anterior (PA) hand/wrist X-ray were taken at the final visit of Core study and at Visit 15/EOS (Month 24) to assess bone age. The change in 2nd metacarpal cortical width at Month 24 relative to the respective Baseline was calculated. If a fracture of the left upper extremity precluded radiographic imaging, (or precluded this X-ray in the Core study) then the right hand was evaluated for this purpose. In this case, an image of the right hand was carried out at both Visit 8 and at Visit 15/EOS (Month 24). The information was used in the assessment of bone density.
Time Frame: Baseline 1 (Visit 1 of the Core Study) and Baseline 2 (Visit 9 of the Extension Study) through Month 24 (Visit 15/Final Extension Visit)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: millimeter (mm)
Arm/Group | Core Treatment Zoledronic Acid | Core Treatment: Placebo
Number analyzed (Participants) | 10 | 15
millimeter (mm)
  2nd metacarpal cortical width change from BL1: number analyzed (Participants) | 6 | 13
  2nd metacarpal cortical width change from BL1 | -0.04 (0.068) | -0.03 (0.054)
  2nd metacarpal cortical width change from BL2 | -0.09 (0.089) | 0.02 (0.063)
Statistical Analysis 1: Comparison: Core Treatment Zoledronic Acid vs Core Treatment: Placebo; 2nd metacarpal cortical width chge from BL1 at Month 24; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.9231, ANCOVA — An analysis of covariance (ANCOVA) model was performed with Core treatment, pooled centers, underlying condition treated with GCs and Core baseline bone age as explanatory variables and pooled centers as random effect; Difference in LS mean = -0.01, 95% CI 2-sided [-0.18 to 0.17]
Statistical Analysis 2: Comparison: Core Treatment Zoledronic Acid vs Core Treatment: Placebo; 2nd metacarpal cortical width chge from BL2 at Month 24; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.2694, ANCOVA — An analysis of covariance (ANCOVA) model was performed with Core treatment, pooled centers, underlying condition treated with GCs and Extension baseline bone age as explanatory variables and pooled centers as random effect; Difference in LS mean = -0.11, 95% CI 2-sided [-0.32 to 0.10]

ADVERSE EVENTS:
Time Frame: Adverse events and serious adverse events were collected for the maximum actual duration of treatment exposure and follow up for a participant per the protocol for approximately 13 months.
Groups:
- Core Treatment Placebo: Twice yearly 0.05 mg/kg (max 5 mg) i.v infusion (at least 30 minutes) of zoledronic acid
Arm/Group | Core Treatment Zoledronic Acid | Core Treatment Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/15
Serious Adverse Events (participants affected / at risk) | 3/10 | 0/15
Other Adverse Events (participants affected / at risk) | 7/10 | 12/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Core Treatment Zoledronic Acid (N=10) | Core Treatment Placebo (N=15)
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Postictal state (Nervous system disorders) | 1 | 0
Status epilepticus (Nervous system disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Core Treatment Zoledronic Acid (N=10) | Core Treatment Placebo (N=15)
Tachycardia (Cardiac disorders) | 1 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 1
Ocular hyperaemia (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 2
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 3
Vomiting (Gastrointestinal disorders) | 2 | 1
Chest pain (General disorders) | 2 | 0
Fatigue (General disorders) | 0 | 3
Infusion site pain (General disorders) | 1 | 0
Pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 2 | 3
Anaphylactic reaction (Immune system disorders) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Candida infection (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 2
Herpes virus infection (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 3
Nasopharyngitis (Infections and infestations) | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 2
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0
Liver function test increased (Investigations) | 0 | 1
Therapeutic agent urine positive (Investigations) | 1 | 0
Vitamin B12 decreased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1
Insulin resistance (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 5
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Trismus (Musculoskeletal and connective tissue disorders) | 0 | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Epileptic aura (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 3 | 2
Postictal state (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 1
Insomnia (Psychiatric disorders) | 0 | 1
Sleep disorder (Psychiatric disorders) | 0 | 2
Suicide attempt (Psychiatric disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Butterfly rash (Skin and subcutaneous tissue disorders) | 1 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 | 0
Tooth extraction (Surgical and medical procedures) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
Secondary hypertension (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-05-18): https://cdn.clinicaltrials.gov/large-docs/00/NCT01197300/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-04): https://cdn.clinicaltrials.gov/large-docs/00/NCT01197300/SAP_001.pdf